CLINICAL TRIAL: NCT02453763
Title: In Vivo Imaging of Therapeutic Electric Current Flow
Acronym: tDCS
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: Arizona State University (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 506-2012-N; 1R21NS081646-01A1 (NIH)
Record Dates: First submitted 2015-05-21; First posted 2015-05-25 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Parkinson Disease; Epilepsy; Alzheimer's Disease; Stroke; Autism; Depression; Schizophrenia
Keywords: Transcranial direct current stimulation; Noninvasive brain stimulation; Brain; Central Nervous System Diseases; Nervous System Diseases; Parkinson disease; Stroke; Epilepsy; Depression; Schizophrenia; Brain imaging; Electrical impedance tomography; Magnetic resonance electrical impedance tomography; Diffusion tensor imaging; Functional magnetic imaging; Rehabilitation
MeSH Terms: conditions — Parkinson Disease; Epilepsy; Alzheimer Disease; Stroke; Autistic Disorder; Depression; Schizophrenia; Central Nervous System Diseases; Nervous System Diseases | interventions — Transcranial Direct Current Stimulation; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Transcranial direct current stimulation: All participants will receive transcranial direct current stimulation and an magnetic resonance imaging (MRI).
  Interventions: Device: Transcranial direct current stimulation; Procedure: MRI

INTERVENTIONS:
Device: Transcranial direct current stimulation — All participants will receive transcranial direct current stimulation. During the MRI images of the head a battery-powered device pulses a small current between a pair of the electrodes which will be immediately followed by more MRI images. The current pulses will be very short and there should be no feeling from the pulses. The entire imaging period will be at most 90 minutes.
  Other Names: Noninvasive Brain Stimulation
Procedure: MRI — All participants will receive an MRI. During the MRI images of the head a battery-powered device pulses a small current between a pair of the electrodes which will be immediately followed by more MRI images. The current pulses will be very short and there should be no feeling from the pulses. The entire imaging period will be at most 90 minutes.
  Other Names: Magnetic Resonance Imaging

SUMMARY:
The purpose of this research study is to measure current flow inside the head using magnetic resonance imaging (MRI). The data from this study will be used to map the current flow caused from the electrical stimulation inside the head. The methods develop will be used to map and better control delivery of the current for electrical stimulation to modify a psychiatric condition such as depression; or other conditions such as epilepsy, Parkinson's disease or autism.

DETAILED DESCRIPTION:
Transcranial direct current stimulation (tDCS) and deep brain stimulation (DBS) are examples of electrical stimulation therapies that are rapidly gaining attention as means of modulating motor function, semantic processing, and executive function. Both therapies have attracted many clinical and experimental studies. tDCS has been found to have both facilitatory and inhibitory effects on the brain depending on stimulation polarity and electrode position. DBS has been thoroughly evaluated clinically for treatment of movement disorders, principally Parkinson's disease, and is extending its reach to include treatment of disorders such as focal dystonia, depression and chronic pain. While still mostly in the experimental stage, tDCS applications and acceptance are growing extremely rapidly.

Although the functional alterations associated with tDCS can be categorized without knowledge of the underlying neurophysiology, an understanding of where externally applied current actually flows in any electrical stimulation technique is crucial as a basis for understanding which brain regions, circuits, or elements are affected by these therapies, and how these changes may occur. Such knowledge will lead to a better understanding of the mechanisms underlying these therapies, and thus to more focused and effective stimulation patterns and locations. Ultimately, this will lead to more efficient and novel clinical applications.

Many studies have simulated the effects of current application in both extra- and intracranial modalities using computer simulation. Simulations will always be limited by errors in interpreting MRI data during segmentation, differences between assumed and actual electrical conductivity values, and mismatches between actual and presumed electrode locations and sizes. Thus, better methods to understand and verify current flow distributions are badly needed.

In this study a recently developed MRI-based phase imaging technique to more directly measure current densities in vivo. Unlike earlier MRI-based methods of measuring electrical current flow, the technique works without requiring subject repositioning. This methods will be validated against high-resolution subject-specific models incorporating many tissue compartments, including anisotropic white matter. Thus, a new direct measurement method against state-of-the-art modeling approaches.

ELIGIBILITY:
Inclusion Criteria:

* right handed (as determined by the Edinburgh battery),
* English as native language.

Exclusion Criteria:

* appreciable deficits in hearing,
* appreciable problems with articulation,
* appreciable accent schizophrenia, bipolar disorder, or major depression,
* any neurological disorder associated with cognitive impairment or neuroanatomic abnormality,
* language-based learning disorder,
* any implanted metal device (precludes use of tDCS), any implanted cardiac pacemaker,
* dementia or mini-mental state exam,
* <24 estimated verbal intelligence,
* <70 active or prior history of seizure disorder, family history of seizure disorder, prescribed seizure inducing medication.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 24 normal adult subjects will be assessed.
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2015-06; Primary Completion 2017-07-06 (Actual); Study Completion 2017-07-06 (Actual)

PRIMARY OUTCOMES:
Magnetic Resonance Imaging (MRI) of therapeutic current flow | Day 1
  The MRI will be used to measure current flow in the brain as a result of therapeutic electrical stimulation techniques by using a recently developed MRI-based phase imaging technique to more directly measure current densities in vivo.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas H Mareci, Ph.D., Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Background] Sadleir RJ, Sajib SZ, Kim HJ, Kwon OI, Woo EJ. Simulations and phantom evaluations of magnetic resonance electrical impedance tomography (MREIT) for breast cancer detection. J Magn Reson. 2013 May;230:40-9. doi: 10.1016/j.jmr.2013.01.009. Epub 2013 Feb 4. PMID 23435264
- [Background] Meng ZJ, Sajib SZ, Chauhan M, Sadleir RJ, Kim HJ, Kwon OI, Woo EJ. Numerical simulations of MREIT conductivity imaging for brain tumor detection. Comput Math Methods Med. 2013;2013:704829. doi: 10.1155/2013/704829. Epub 2013 Apr 29. PMID 23737862
- [Background] DeMarse TB, Carney PR. Augmentation of cognitive function in epilepsy. Front Syst Neurosci. 2014 Aug 14;8:147. doi: 10.3389/fnsys.2014.00147. eCollection 2014. No abstract available. PMID 25177279
- [Result] Sadleir RJ, Vannorsdall TD, Schretlen DJ, Gordon B. Target optimization in transcranial direct current stimulation. Front Psychiatry. 2012 Oct 17;3:90. doi: 10.3389/fpsyt.2012.00090. eCollection 2012. PMID 23087654